CLINICAL TRIAL: NCT04781491
Title: Effects of Nature and Forest Therapy in Patients With Metabolic Syndrome and Cardiovascular Risk Factors - a Randomized Controlled Trial
Brief Title: Effects of Nature and Forest Therapy in Patients With Metabolic Syndrome and Cardiovascular Risk Factors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Andreas Michalsen, Prof.Dr.med, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Wald
Record Dates: First submitted 2021-02-23; First posted 2021-03-04 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Metabolic Syndrome, Protection Against
Keywords: Forest Therapy; Forest Bathing; Shinrin Yoku; Metabolic Syndrome; Cardiovascular Risks
MeSH Terms: conditions — Metabolic Syndrome | interventions — Forest Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Forest Therapy (Düppeler Forst - Berlin-Wannsee) (Experimental): Subjects receive a 90-minute Forest Therapy session once per week for 8 weeks with a licensed nature therapist, who explains exercises on perceiving nature and the connection between nature and health.
  Interventions: Behavioral: Forest Therapy (Düppeler Forst - Berlin-Wannsee)
- Waiting list (No Intervention): Subjects don't receive any therapy but are offered the same treatment after trial is finished.

INTERVENTIONS:
Behavioral: Forest Therapy (Düppeler Forst - Berlin-Wannsee) — Forest Therapy means mindful visits in nature, actively perceiving the flora and fauna
  Arms: Forest Therapy (Düppeler Forst - Berlin-Wannsee)

SUMMARY:
The aim of this study is to investigate the effects of regular forest therapy under guidance of a licensed nature therapist on patients with metabolic syndrome and cardiovascular risks

DETAILED DESCRIPTION:
It is assumed that nature and forest experience has sustainable benefits for the physical and mental health of individuals with metabolic syndrome and cardiovascular risk profile. Especially co-therapeutic effects in terms of resilience and salutogenesis might effectively and sustainably promoted by nature and forest therapy.

The main objective of this study is to measure the effects of nature and forest therapy in subjects with manifest metabolic syndrome and cardiovascular risk factors. The intervention is a stay in the nature of the Düppeler Forest (Berlin-Wannsee) under the guidance of trained nature guides (90 minutes, 1x/week over 2 months), who teach exercises on the perception of nature and the connection between nature and health, movement and mindfulness. Subjects are also motivated to experience forest nature as regularly as possible (recommended ≥ 30 minutes daily). Participants of the control group will be offered a later participation in the therapy program after completion of the last study visit after 4 months (waiting list control group).

ELIGIBILITY:
Inclusion Criteria:

* Definition of Metabolic Syndrome according to the International Diabetes Foundation (IDF):
* waist circumference: at least 94 cm for men, at least 80 cm for women
* plus at least two of the following risk factors:
* fasting blood glucose levels of > 100 mg/dl (> 5.6 mmol/l) measured in blood plasma or diagnosed diabetes mellitus
* elevated triglycerides > 150 mg/dl (> 1.7 mmol/l) or therapy already initiated to lower triglycerides
* low HDL cholesterol: < 40 mg/dl (< 1.05 mmol/l) in men and < 50 mg/dl (< 1.25 mmol/l) in women or already initiated therapy to increase HDL
* Hypertension (from > 130 mmHg systolic and > 85 mmHg diastolic) or already treated hypertension

Exclusion Criteria:

* Serious acute or chronic illnesses
* Immobility or limitation of mobility due to orthopedic, neurological or other medical cause
* Participation in another study
* Serious mental illness
* Pregnancy and lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-06-27 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
• Final sum score of cardiovascular risk profile (overweight, blood pressure, blood lipids, blood glucose) according to Wiley/Carrington | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks

SECONDARY OUTCOMES:
• Perceived Stress Scale (PSS) | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks]
  Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived•stress. Higher score meaning more stress
• Short Form 12 Health Survey (SF-12) | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks]
  The Short Form (12) Health Survey is a 12-item, patient-reported survey of patient health.The World Health Organisation- Five Well-Being Index (WHO-5) is a short self-reported measure of current mental wellbeing. score ranging from 0-5 for each question, lower score meaning a better outcome.
• Physical complaints (B-LR - Beschwerden-Liste) | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks]
  the Complaints List - (B-LR) is a self-assessment procedure for recording subjective impairment due to physical or general complaints, covering the entire spectrum from no complaints to severe impairment. Two parallel forms (B-LR and B-LR') are available, each consisting of 20 items, lower score meaning a better outcome
• Flourishing Scale (FS-D) | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks]
  The Flourishing Scale is a brief 8-item summary measure of the respondent's self-perceived success in important areas such as relationships, self-esteem, purpose, and optimism. The scale provides a single psychological well-being score, ranging from 8-56, higher score meaning a better outcome
• Hospital Anxiety and Depression Scale (HADS) | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks]
• Mindfulness (Freiburger Fragebogen zur Achtsamkeit, FFA) | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks]
  Assessing full scale, range 0-56, higher score meaning a better outcome
• General Self-Efficacy Short Scale (ASKU-Allgemeine Selbstwirksamkeit Kurzskala) | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks]
  Measurement instrument for recording subjective competence expectations. Scale ranging from 1-5, higher score meaning a better outcome
• International Physical Activity Questionnaire (IPAQ) | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks]
  The 31-item long form and the 9-item short form assess time spent on different activities. The short form records four types of physical activity: vigorous activity such as aerobics; moderate-intensity activity such as leisure cycling; walking, and sitting.
  MET minutes represent the amount of energy expended carrying out physical activity. To get a continuous variable score from the IPAQ (MET minutes a week) we will consider walking to be 3.3 METS, moderate physical activity to be 4 METS and vigorous physical activity to be 8 METS; higher score meaning better outcome; range 0 to around 3000 MET minutes a week
• Weekly query of the exercise practice by means of (online) diary | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks]
Subjective Vitality Scale state (SVS-G state) | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks
  Assessing full scale, range 1-80, higher score meaning a better outcome
Perceived Benefits of Nature Questionnaire (PBNQ) | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks
  Assessing full scale, range 1-7, lower score meaning a better outcome
Profile of Mood States (POMS) | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks

OTHER OUTCOMES:
- Blood count | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks]
  Laboratory parameters
- Blood lipids (total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides) | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks]
  Laboratory parameters
- Parameters of glucose metabolism (insulin, glucose, HbA1C, insulin sensitivity) | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks]
  Laboratory parameters will be combined to report Diabetes status
- liver function (GOT, GPT, GGT) | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks]
  Laboratory parameters
- Inflammation: hs-CRP, IL-6 | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks]
  Laboratory parameters
- IFN-gamma, tumor necrosis factor alpha | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks]
  Laboratory parameters
- uric acid | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks]
  Laboratory parameters
- Lymphocyte populations: T cells (CD3), B cells (CD19), NK cells (CD16). | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks]
  Laboratory parameters
- T cell subpopulations: T helper cells (CD4), cytotoxic T cells (CD8), CD4/CD8 ratio. | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks]
  Laboratory parameters
- ferritin | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks]
  Laboratory parameters
- cumulative steroid hormone concentration of the last 2 months in a hair strand | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks]
  Laboratory parameters
• Apparatus parameters | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks]
  * Body weight
  * abdominal girth
  * blood pressure measurement (24h) will be combined to report metabolic syndrome
• Qualitative evaluation (focus group interviews) | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks]
  - Semi-structured interviews and focus group discussions with 16 subjects of the intervention group.
• Heart rate variability and other parameters | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks]
  - Digital tracking using "wearables": parameters of stress levels and activity and sleep patterns are measured objectively using a smartwatch (fitbit). Heart rate variability (RMSSD), pulse, activity duration, type, and intensity as well as sleep duration, sleep phases, steps, and calorie consumption are recorded. The aim is to test whether the activity and pulse tracking data provide information about the variance in quality of life data. Will be combined to report quality of life.
- bioelectrical impedance analysis (BIA) | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks]
  Estimation of the body composition via bio-electrical impedance analysis (muscle mass in kg)
Heart Rate (HR) | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  24h measuring by smartwatch
Heart Rate Variability (HRV) | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  24h measuring by smartwatch
Interbeat Interval (IBI) | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  24h measuring by smartwatch
Number of steps | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  24h measuring by smartwatch

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Michalsen, Prof. Dr., Principal Investigator — Charité Hochschulambulanz für Naturheilkunde am Immanuel Krankenhaus
Locations (1):
- Charité Hochschulambulanz für Naturheilkunde am Immanuel Krankenhaus, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes